CLINICAL TRIAL: NCT05157438
Title: Comparative Evaluation of The Effect of Virtual Reality and Screen Programs on Children's Dental Anxiety, Pain and Behavior: A Randomized Cross-Over Clinical Trial
Brief Title: Effect of VR vs Screens on Children's Dental Anxiety, Pain and Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amal Salem Yousry Mahrouse, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VR in Child Anxiety
Record Dates: First submitted 2021-11-11; First posted 2021-12-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dental Anxiety
Keywords: virtual reality
MeSH Terms: interventions — Tablets; Television

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (virtual reality group) (Experimental): The virtual reality device is a 3D head-mounted display which provides a wide field of view and a high-resolution visual display, the system consists of head mounted glasses, a compatible smartphone and headphones. This technology creates a computer stimulated virtual environment.
  Interventions: Behavioral: virtual reality device
- Group II (screen program group). (Active Comparator): the screens shows such as cartoons, animation movies or recorded video games are used for distraction during dental treatments. They could be seen on tablets, iPads or LCD screen.
  Interventions: Behavioral: screen programs

INTERVENTIONS:
Behavioral: virtual reality device — The virtual reality device is a 3D head-mounted display which provides a wide field of view and a high-resolution visual display, it has been used to manage cases of phobia and extreme fear through the use of exposure-based treatment programs. The virtual reality system consists of head mounted glasses, a compatible smartphone and headphones. This technology creates a computer stimulated virtual environment into which the child can be entirely immersed. It works to distract the brain from the painful procedure and reduce the perception of pain stimuli
  Arms: Group I (virtual reality group)
Behavioral: screen programs — the screens are used for distraction during dental treatments. they could be on tablets, iPads or televisions.
  Other Names: tablets, televisions
  Arms: Group II (screen program group).

SUMMARY:
Virtual reality distraction is intended to reduce the pain experience by distracting the patient attention from the pain stimulating procedure. Then, it breaks the cycle of negative experiences by improving the dental experience. The study's aim is to compare the effect of virtual reality to the effect of screen programs on dental anxiety, pain and behavior at different time points among children undergoing dental treatment under local anesthesia. The null hypothesis assumes that virtual reality has no effect on reducing the children's pain or anxiety and there is no difference between virtual reality and screen programs in improving the children's behavior and dental experience. The study's design is a cross-over, split mouth trial in which each patient will have similar dental treatments on each side, but with different distraction techniques.

DETAILED DESCRIPTION:
Most of dental procedures are accompanied by pain and discomfort which subsequently adversely affect the patient's cooperation and willingness to complete or undergo the procedures. This negative behavior compromises the efficiency and quality of the delivered dental treatment, to the extent that it may not be completed. Therefore, behavior management techniques have been introduced to the field of pediatric dentistry to effectively manage the child anxiety and improve the child's experience in dental office to establish a positive child-dentist relationship. The virtual reality (VR) is considered a behavior management technique as well as a distraction tool, as it modifies the child's attitude. Thus, it can be used in the dental practice to help the dentist to control the child during the treatment procedure. The study's design is a cross-over, split mouth trial in which the procedure is planned to be on three visits, as the following: baseline visit (v0) for diagnosis, examination and inclusion, first visit (v1) and second visit (v2) for treatment sessions. A follow up visit (v3) may be needed for younger patients who need space maintenance for the extraction site. allocated and randomized equally into two groups according to the intervention assigned in the first treatment session: Group I (virtual reality group) and Group II (screen program group). In both groups, children will be allowed to choose an animation or cartoon from a list pre-prepared by the investigator in order to watch a show of their own choice, to augment the effect of distraction. Both groups will be managed and operated by the same operator who is the research investigator. Treatments were completed in two separate sessions, two weeks apart as a washout period, to avoid any carry-over effect. Each patient will have two teeth extracted, one on each side, on two successive visits, with two weeks apart as a washout period. The required sample size was calculated using the IBMª SPSSª Sample Powerª version 3.0.1 (IBMª Corp., Armonk, NY, USA). Subjects will be recruited from the outpatient clinic in Pediatric Dentistry and Dental Public health Department. Faculty of Dentistry, Cairo University, Egypt. Patients will be screened by the research investigator until the target population is achieved. The outcome data and results will be independently collected from each participant by the researcher, examined, organized and analyzed under the supervision of the assistant supervisor. Any missing data will be revised and handled with the best techniques according to the type of data missed. All data will be entered and stored on a secured personal computer in coded and password locked files. Backup of data on an external hard disc in order to prevent any data loss. Results will be statistically analyzed by using statistical package of social sciences (SPSS 26.0, IBM/SPSS Inc., Chicago, IL). There are two types of statistical methods Descriptive statistics and Analytical or inferential statistics. In this study, no data monitoring committee will be needed since it is a study with known minimal risks. The Main Supervisor will monitor this study. Auditing will be done by the main and co-supervisors to assure quality of the research methods, restorative technique and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children between 5-7 years old age.
* Both genders.
* First dental visit
* Positive and definitely positive behavior according to Frankel behavior scale.
* Two or more badly decayed primary maxillary first molars beyond repair and need to be extracted.
* Systemically and mentally healthy.

Exclusion Criteria:

* History of systemic or mental conditions.
* Special health care needs who require pharmacological management prior to dental treatment.
* Acute dental pain or trauma.
* Extremely uncooperative children who require being treated under general anesthesia, negative and definitely negative according to Frankel behavior scale

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
RMS Pictorial Scale: A scale to assess the change in dental anxiety through the dental procedure | The dental anxiety is measured during same single visit. There is no follow up and no specific time duration for the visit. Pre-operative anxiety: before administration of local anesthesia and Post-operative anxiety: after dental extraction.
  The scale consists of row of 5 photographs of a child showing 5 different faces ranging from happy to very unhappy. The child is asked to choose the face that looks like what they feel at the moment. The score is recorded by giving value of 1 to happy and value of 5 to very unhappy. The RMS-pictorial scale is chosen for simple and easy for the child to understand, has 2 sets of photographs for boys and for girls, which gives efficient evaluation of dental anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Amal S Abdelatty, Masters, Principal Investigator — Cairo University; Cairo University, Study Chair — 11 El-Saraya St. - Manial - Cairo
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Nunna M, Dasaraju RK, Kamatham R, Mallineni SK, Nuvvula S. Comparative evaluation of virtual reality distraction and counter-stimulation on dental anxiety and pain perception in children. J Dent Anesth Pain Med. 2019 Oct;19(5):277-288. doi: 10.17245/jdapm.2019.19.5.277. Epub 2019 Oct 30. PMID 31723668
- [Background] Rao DG, Havale R, Nagaraj M, Karobari NM, Latha AM, Tharay N, Shrutha SP. Assessment of Efficacy of Virtual Reality Distraction in Reducing Pain Perception and Anxiety in Children Aged 6-10 Years: A Behavioral Interventional Study. Int J Clin Pediatr Dent. 2019 Nov-Dec;12(6):510-513. doi: 10.5005/jp-journals-10005-1694. PMID 32440065
- [Background] Tanja-Dijkstra K, Pahl S, White MP, Andrade J, Qian C, Bruce M, May J, Moles DR. Improving dental experiences by using virtual reality distraction: a simulation study. PLoS One. 2014 Mar 12;9(3):e91276. doi: 10.1371/journal.pone.0091276. eCollection 2014. PMID 24621518
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Nuvvula S, Alahari S, Kamatham R, Challa RR. Effect of audiovisual distraction with 3D video glasses on dental anxiety of children experiencing administration of local analgesia: a randomised clinical trial. Eur Arch Paediatr Dent. 2015 Feb;16(1):43-50. doi: 10.1007/s40368-014-0145-9. Epub 2014 Sep 26. PMID 25256207
- [Background] Niharika P, Reddy NV, Srujana P, Srikanth K, Daneswari V, Geetha KS. Effects of distraction using virtual reality technology on pain perception and anxiety levels in children during pulp therapy of primary molars. J Indian Soc Pedod Prev Dent. 2018 Oct-Dec;36(4):364-369. doi: 10.4103/JISPPD.JISPPD_1158_17. PMID 30324926